CLINICAL TRIAL: NCT05702398
Title: Pilot Trial of Supplemental Vitamin A and Nicotinamide and Levels of Blood Vitamin A and Nicotinamide
Brief Title: Pilot Trial of Supplemental Vitamin A and Nicotinamide
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19792
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-12

CONDITIONS: Skin Cancer; Kidney Transplant Recipients
MeSH Terms: conditions — Skin Neoplasms | interventions — Vitamin A; Niacinamide; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin A & Nicotinamide (Experimental): 1,000 μg retinyl palmitate and 500 mg NAM twice a day
  Interventions: Drug: Vitamin A; Drug: Nicotinamide
- Placebo (Placebo Comparator): Identical placebo pills twice a day
  Interventions: Other: Other: Placebo

INTERVENTIONS:
Drug: Vitamin A — 1,000 μg retinyl palmitate twice a day for 6 months
  Arms: Vitamin A & Nicotinamide
Drug: Nicotinamide — 500 mg NAM twice a day for 6 months
  Other Names: Niacin (Vitamin B3)
  Arms: Vitamin A & Nicotinamide
Other: Other: Placebo — Identical placebo pills twice a day
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the feasibility and safety of oral nicotinamide (NAM; a derivative of vitamin B3 [niacin]) and vitamin A in a high-risk population of kidney transplant recipients with a history of skin cancer to generate preliminary data for future cancer prevention clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater;
* Either History of 2 or more histologically confirmed invasive cutaneous SCCs in the past 2 years or
* At least one previously billed Healthcare Common Procedure Coding System code 17004 (destruction of 15 or more benign or premalignant lesions of the integumentary system);
* Understands, reads, and writes English proficiently.

Exclusion Criteria:

* Liver disease;
* Active peptic ulcer disease;
* Recent myocardial infarction;
* Hypotension;
* Internal malignancy within past 5 years;
* Renal impairment with eGFR<15 mL/min/1.73 m2;
* Being unable for follow up due to social reasons;
* Gorlin's syndrome or other genetic skin cancer syndrome;
* Huge number of current skin cancers;
* Metastatic SCC or invasive melanoma within the past 5 years;
* Pregnancy or lactation;
* Need for ongoing carbamazepine use (which could have a possible interaction with NAM);
* Use of acitretin or other oral retinoids within the past 6 months;
* Use of supplemental NAM, niacin, vitamin A, or beta carotene within the past 6 months;
* Field treatment for actinic keratoses (AKs) within the previous 4 weeks;
* Use of topical steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of Blood Vitamin A and Nicotinamide Levels | 6 months

IPD SHARING:
Plan to Share IPD: Undecided